CLINICAL TRIAL: NCT05216666
Title: Abductor Insufficiency After Total Hip Arthroplasty; Risk Factors and Diagnosis
Brief Title: The Role of Surgical Approach on Residual Limping After Total Hip Arthroplasty
Acronym: HSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Georgios Tsikandylakis, MD PhD, Senior consultant in orthopaedic surgery, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 277461
Record Dates: First submitted 2022-01-15; First posted 2022-01-31 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hip Osteoarthritis; Muscle Weakness; Muscle Atrophy; Muscle Injury; Arthroplasty Complications
Keywords: abductor; approach; limp; Trendelenburg; gluteus medius
MeSH Terms: conditions — Osteoarthritis, Hip; Muscle Weakness; Muscular Atrophy; Intermittent Claudication

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral approach (Active Comparator): 290 participants receive their hip prosthesis through a lateral approach. The anterior third of m. gluteus medius along with the corresponding part of m. vastus lateralis are detached from the greater trochanter and the anterior capsule is excised for the exposure of the hip joint. After implant insertion, the gluteus medius is reinserted into the greater trochanter with non-absorbable sutures. Participants are followed at three and 12 months by a physiotherapist.
  Interventions: Procedure: Lateral approach
- Posterior approach (Active Comparator): 290 participants receive their hip prosthesis through a posterior approach. The m. piriformis gemelli and obturator internus are detached from the greater trochanter and the posterior capsule is incised for the exposure of the hip joint. After implant insertion, the posterior capsule as well as m piriformis and the external rotators are reinserted into the greater trochanter with non-absorbable sutures. Participants are followed at three and 12 months by a physiotherapist.
  Interventions: Procedure: Posterior approach

INTERVENTIONS:
Procedure: Lateral approach — Total hip arthroplasty performed through a lateral surgical approach (Gammer)
  Other Names: Gammer approach
  Arms: Lateral approach
Procedure: Posterior approach — Total hip arthroplasty performed through a posterior surgical approach (Moore)
  Other Names: Moore approach
  Arms: Posterior approach

SUMMARY:
Residual limping after total hip arthroplasty is empirically associated with the use of lateral approach but has been reported in litterature even with the use of posterior approach. The purpose of this clinical trial is to compare the risk of residual limping one year after total hip arthropasty between lateral and posterior approach.

DETAILED DESCRIPTION:
The use of lateral approach has been empirically associated with increased risk of abductor insufficiency and limping after total hip arthroplasty compared with the posterior approach. However lateral approach remains a widespread technik because it provides a decreased risk of dislocation. In litterature, gluteus medius insufficiency has been reported even when the posterior approach has been used. In the early stage of postperative relhabilitation it is difficult to distinguish between between limping that resolves after abductor training and limping due to abductor injury/avulsion that is resistent to physiotherapy. The purpose of this randomized controlled trial is to compare the risk of persistent limping one year after total hip arthtoplasty between lateral and posterior approach and to identify patient-related risk factors for limping. Moreover it will validate ultra sound (U/S), magnetic resonance imaging (MRI) of the hip and gait analysis as diagnostic tools for early detection of limping that is going to persist one year after total hip arthroplasty.

580 patients will hip osteoarthritis be randomised to receive their total hip arthroplasty through an either lateral of posterior approach and will be followed at one year with physical examination (Trendelenburg sign) and patient.-reported outcome measures. Patients with a positive Trendelenburg sign at 3 months will undergo U/S and MRI examination as well as gait analysis and reassessed at one year with physical examination. The first 40 patients with negative Trendelenburg sign at 3 months will also undergo U/S, MRI and gait analysis. The specificity and sensitivity of U/S, MRI and gait analysis for positiv Trendelenburg sign will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral osteoarthritis of the hip scheduled for total hip arthroplasty.
* Ability to understand and write swedish.

Exclusion Criteria:

* Impaired funktion of the contralateral hip or knees causing limping.
* Neuromuscular diseases
* Postoperative leg length discrepancy excceding 1 cm
* Postoperative discrepancy in femoral offset exceeding 25% of the femoral offset of the contralateral hip.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Trendelenburg sign as binary variable (positive/negative) | At 12 months after intervention
  Trendelenburg sign negative if the pelvis remains horisontal while standing only on the operated leg with both arms in anatomical postion. If the pelvismcannot be kept horisontal and tilts towards the kontralateral hip the Trendelenburgs sign is regarded as positive.

SECONDARY OUTCOMES:
Dislocation | Within 12 months from intervention
  Incidens of postoperative dislocation
Intraoperative blood loss | Intraoperative
  Bleeding during total hip arthroplasty measured in ml
Periprosthetic infection | Within 12 months from intervention
  Incidens of deep surgical wound infection
Oxford Hip Score | At 3 months after intervention
  Patient-reported hip function measured in a scale of 0-48
Oxford Hip Score | At 12 months after intervention
  Patient-reported hip function measured in a scale of 0-48
Euroqol 5 dimension 5 level index (EQ5D-5L) | At 3 months after intervention
  Patient-reported health-related quality of life measured with the swedish version of euroqol 5 dimension 5 level index 0-1
Euroqol 5 dimension 5 level index (EQ5D-5L) | At 12 months after intervention
  Patient-reported health-related quality of life measured with the swedish version of euroqol 5 dimension 5 level index 0-1
Euroqol visual analog scale (EQVAS) | At 3 months after intervention
  Patient-reported health-related quality of life measured with the euroqol visual analog scale 0-100
Euroqol visual analog scale (EQVAS) | At 12 months after intervention
  Patient-reported health-related quality of life measured with the euroqol visual analog scale 0-100
University of California Activity Level (UCLA) | At 3 months after intervention
  Patient-reported acivity level measured with the University of California Level of Acivity rank scale 0-10
University of California Activity Level (UCLA) | At 12 months after intervention
  Patient-reported acivity level measured with the University of California Level of Acivity rank scale 0-10
Gluteus medius avulsion in ultrasound | At 3 months after intervention
  The proportion avulsed gluteus medius tendon in relation to the whole tendon attachment in a scale of 0 (no avulsion) to 1 (total avulsion). Measured with ultrasound
Gluteus medius atrophy in Magnetic Resonance Imaging | At 3 months after intervention
  The area of gluteus medius muscle in the operated side divided by the area of the gluteus medius muscle in the healthy side as shown in magnetic resonance imaging in a scale of 0 (complete atrophy) to 1 (no atrophy)
Hip abuction torque | At 3 months after intervention
  Hip abuction torque measured in Nm/Kg with gate analysis
Trendelenburg sign as binary variable (positive/negative) | At 3 months after intervention
  Trendelenburg sign negative if the pelvis remains horisontal while standing only on the operated leg with both arms in anatomical postion. If the pelvismcannot be kept horisontal and tilts towards the kontralateral hip the Trendelenburgs sign is regarded as positive.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Tsikandylakis, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hailer NP, Weiss RJ, Stark A, Karrholm J. The risk of revision due to dislocation after total hip arthroplasty depends on surgical approach, femoral head size, sex, and primary diagnosis. An analysis of 78,098 operations in the Swedish Hip Arthroplasty Register. Acta Orthop. 2012 Oct;83(5):442-8. doi: 10.3109/17453674.2012.733919. Epub 2012 Oct 8. PMID 23039167
- [Background] Zijlstra WP, De Hartog B, Van Steenbergen LN, Scheurs BW, Nelissen RGHH. Effect of femoral head size and surgical approach on risk of revision for dislocation after total hip arthroplasty. Acta Orthop. 2017 Aug;88(4):395-401. doi: 10.1080/17453674.2017.1317515. Epub 2017 Apr 25. PMID 28440704
- [Background] Skoogh O, Tsikandylakis G, Mohaddes M, Nemes S, Odin D, Grant P, Rolfson O. Contemporary posterior surgical approach in total hip replacement: still more reoperations due to dislocation compared with direct lateral approach? An observational study of the Swedish Hip Arthroplasty Register including 156,979 hips. Acta Orthop. 2019 Oct;90(5):411-416. doi: 10.1080/17453674.2019.1610269. Epub 2019 May 7. PMID 31060427
- [Background] Moerman S, Mathijssen NMC, Tuinebreijer WE, Vochteloo AJH, Nelissen RGHH. Hemiarthroplasty and total hip arthroplasty in 30,830 patients with hip fractures: data from the Dutch Arthroplasty Register on revision and risk factors for revision. Acta Orthop. 2018 Oct;89(5):509-514. doi: 10.1080/17453674.2018.1499069. Epub 2018 Aug 6. PMID 30080985
- [Background] Whiteside LA, Roy ME. Incidence and treatment of abductor deficiency during total hip arthroplasty using the posterior approach: repair with direct suture technique and gluteus maximus flap transfer. Bone Joint J. 2019 Jun;101-B(6_Supple_B):116-122. doi: 10.1302/0301-620X.101B6.BJJ-2018-1511.R1. PMID 31146555
- [Background] Ewen AM, Stewart S, St Clair Gibson A, Kashyap SN, Caplan N. Post-operative gait analysis in total hip replacement patients-a review of current literature and meta-analysis. Gait Posture. 2012 May;36(1):1-6. doi: 10.1016/j.gaitpost.2011.12.024. Epub 2012 Mar 10. PMID 22410129